CLINICAL TRIAL: NCT00667693
Title: A Randomized Comparison Between the Pentax AWS Video Laryngoscope and the Macintosh Laryngoscope
Brief Title: Pentax Airway Scope (AWS) Intubation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 08-046
Record Dates: First submitted 2008-04-24; First posted 2008-04-28 (Estimated); Results first posted 2016-10-31 (Estimated); Last update posted 2018-07-24 (Actual); Status verified 2018-07

CONDITIONS: Obesity
Keywords: intubation; obese
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Macintosh laryngoscope (Active Comparator): Intubation with a Macintosh laryngoscope
  Interventions: Device: Macintosh laryngoscope
- Pentax AWS (Active Comparator): Intubation with a Pentax AWS
  Interventions: Device: Pentax AWS

INTERVENTIONS:
Device: Macintosh laryngoscope — Intubation with Macintosh laryngoscope
  Arms: Macintosh laryngoscope
Device: Pentax AWS — Intubation with Pentax AWS
  Arms: Pentax AWS

SUMMARY:
This study will compare the Macintosh laryngoscope with the Pentax. The Pentax AWS is a novel airway management device that is designed to facilitate laryngoscopy and endotracheal intubation.

DETAILED DESCRIPTION:
100 obese patients (BMI 30 to 50) requiring orotracheal intubation for elective surgery will be randomly allocated to intubation with either a conventional Macintosh laryngoscope or with the Pentax AWS. Our study hypothesis is that use of Pentax AWS will make tracheal intubation easier to perform in the obese surgical patient (BMI 30 to 50), as evidenced by the time to complete the intubation process as well as an "Ease of Use" visual analog score (VAS) measure.

ELIGIBILITY:
Inclusion Criteria:

* subject is at least 18 years old
* BMI between 30 and 50
* scheduled for elective surgery requiring orotracheal intubation

Exclusion Criteria:

* a known difficult airway
* loose teeth
* subject pregnancy
* rapid sequence induction required
* subject is unable to give consent
* anesthesiologist considered use of the Pentax AWS to be contraindicated
* special endotracheal tube (ETT) is needed for the case.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2008-02; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel I Sessler, MD, Study Chair — The Cleveland Clinic; John Doyle, MD, PhD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Macintosh: Intubation with a Macintosh laryngoscope
  Macintosh intubation: Macintosh intubation
- Pentax: intubation with a the Pentax AWS
  Pentax AWS: Intubation with Pentax AWS
Period: Overall Study
Arm/Group | Macintosh | Pentax
Started | 49 | 52
Completed | 49 | 50
Not Completed | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Macintosh | Pentax | Total
Number analyzed (Participants) | 49 | 50 | 99
Age, Continuous [Mean (Standard Deviation); unit: years] | 49 (14) | 50 (12) | 49 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 39 | 78
  Male | 10 | 11 | 21
Region of Enrollment [Number; unit: participants]
  United States | 49 | 50 | 99
ASA status [Number; unit: participants] — American Society of Anesthesiology (ASA) physical status classification system
  participants
    II: mild systemic disease | 7 | 15 | 22
    III: severe systemic disease | 40 | 32 | 72
    IV: severe systemic disease that threats to life | 2 | 3 | 5
Mallampati score [Number; unit: participants]
  1: Soft palate, uvula, fauces, pillars visible | 14 | 21 | 35
  2: Soft palate, uvula, fauces visible | 21 | 18 | 39
  3: Soft palate, base of uvula visible | 13 | 7 | 20
  4: Only hard palate visible | 0 | 4 | 4

OUTCOME MEASURES:

1. Primary Outcome: Time to Intubation
Description: time between sufficient muscle relaxant and placement of intubation tube
Time Frame: time between sufficient muscle relaxant and placement of intubation tube, up to 100 seconds
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | Macintosh | Pentax
Number analyzed (Participants) | 49 | 50
seconds | 26 [22 to 29] | 38 [31 to 50]
Statistical Analysis 1: Comparison: Macintosh vs Pentax; Test type: Superiority or Other; p < 0.001, Regression, Cox; Hazard Ratio (HR) = 0.35, 95% CI 2-sided [0.23 to 0.55]

2. Secondary Outcome: Ease of Intubation
Description: Ease of intubation was recorded by the operator immediately after intubation on a 100 mm visual analog scale (VAS). The score ranges from 0 to 100. A higher score indicates more difficulty in intubation
Time Frame: From the start of intubation until 24 hours after surgery
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Macintosh | Pentax
Number analyzed (Participants) | 49 | 50
units on a scale | 40 (28) | 52 (31)

3. Secondary Outcome: Successful Intubation on the First Attempt
Description: The count number of successful intubation on the first attempt
Time Frame: From the start of intubation until 24 hours after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Macintosh | Pentax
Number analyzed (Participants) | 49 | 50
Participants | 45 | 43

4. Secondary Outcome: The Number of Patients With Different Number of Intubation Attempts
Description: We summarized the number of patients with one, two or three intubation attempts.
Time Frame: From the start of intubation until 24 hours after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Macintosh | Pentax
Number analyzed (Participants) | 49 | 50
Participants
  one attempt | 45 | 44
  two attempts | 4 | 3
  three attempts | 0 | 3

5. Secondary Outcome: The Number of Patients With Bleeding
Time Frame: From the start of intubation until 24 hours after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Macintosh | Pentax
Number analyzed (Participants) | 49 | 50
Participants | 0 | 2

ADVERSE EVENTS:
Time Frame: From the start of intubation until 24 hours after surgery
Arm/Group | Macintosh | Pentax
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/50
Other Adverse Events (participants affected / at risk) | 0/49 | 0/50

LIMITATIONS AND CAVEATS:
It focused on obese patients; did not include patients with a history of difficult intubation; protocol did not include use of adjunctive devices; was impossible to blind the operator to the device being used; only the Mallampati score was recorded

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes